CLINICAL TRIAL: NCT06756412
Title: Investigation of the Efficacy of an Exercise Regimen Following Arthrocentesis in the Management of Temporomandibular Disorders
Brief Title: The Effects of an Exercise Regimen Following TMJ Arthrocentesis
Acronym: ExeTMJArthro
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Aras Erdil, Assistant Professor Doctor, Tokat Gaziosmanpasa University
Other Study IDs: UsakU
Record Dates: First submitted 2024-12-25; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders; Arthrocentesis; Temporomandibular joint; Exercise Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arthrocentesis Group: Patients with arthralgia and limited mouth opening at least 3 moths, if volunteered, will be enrolled to this group. The patients will undertake a TMJ arthrocentesis, will be recommended behavioural modifications and diet alterations.
  Interventions: Procedure: Temporomandibular Joint Arthrocentesis
- Self-Exercise Following TMJ Arthrocentesis: Patients with arthralgia and limited mouth opening at least 3 moths will be enrolled to this group. The patients, if volunteered, will undertake a TMJ arthrocentesis, will be recommended behavioural modifications and diet alterations. Following the arthrocentesis procedure, the patients will be instructed an exercise regimen adopted from the current literature, and asked to perform the regimen for postoperative six weeks.
  Interventions: Procedure: Self Exercise Following Arthrocentesis

INTERVENTIONS:
Procedure: Temporomandibular Joint Arthrocentesis — The symptomatic temporomandibular joint (TMJ), either right or left, will be anesthetized using an auriculotemporal nerve block and intracapsular anesthesia. The arthrocentesis procedure will be performed using the double-puncture technique. A 21-gauge needle will be inserted into the posterior region of the joint capsule, targeting the upper joint compartment at a point located 10 mm anterior to the tragus. A second 21-gauge needle will be introduced into the anterior region of the joint capsule, also targeting the upper compartment, at a point located 20 mm anterior to the tragus. The upper joint compartment will then be irrigated with a minimum of 200 mL of saline solution through one of the needles.
  Groups: Arthrocentesis Group
Procedure: Self Exercise Following Arthrocentesis — Following the arthrocentesis procedure described for the other study group, patients will undergo a standardized exercise regimen based on established literature. The regimen includes two sets of movements. The first set involves freely opening the jaw, shifting it right, left, and forward, and repeating these movements while applying finger resistance-closing the mouth against the pressure or forcing the jaw open with the fingers. Each movement will last 10 seconds and be performed 10 times daily. The second set aims to improve the mandibular condyle-articular disc relationship. Patients will open their mouth as wide as possible, advance their lower jaw fully, and close their teeth in an edge-to-edge position. These movements will be performed three times daily for 5 minutes after meals.
  Groups: Self-Exercise Following TMJ Arthrocentesis

SUMMARY:
The goal of this study is to evaluate the short- and long-term effects of a self-administered exercise program on pain levels, jaw movement range, and jaw function in patients with temporomandibular joint (TMJ) disorders. The main question it aims to answer is:

Does adding a self-administered exercise program to arthrocentesis improve pain, mouth opening, and jaw function compared to arthrocentesis alone in patients with TMJ disorders?

Participants with acute or chronic TMJ pain lasting at least three months and limited mouth opening will undergo arthrocentesis, with one group also following an exercise regimen. Outcomes will be assessed over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Limited mouth opening (<35mm) and joint pain complaints according to the DC/TMD examination form,
* Pain complaints for 3 months or longer,
* Able to understand Turkish in spoken and written language,
* Patients who can read the written consent form and give signed consent will be included in the study.

Exclusion Criteria:

* Those with serious neurological disorders,
* Those with autoimmune disorders involving muscles or joints,
* Those with a history of alcoholism,
* Patients diagnosed with malignancy,
* Patients who have previously undergone surgery or radiotherapy in the head and neck region,
* Those with other TMD diagnoses that do not cause restriction or pain in mouth opening,
* Those who have received other treatments for the neck or TMJ regions in the last 3 months,
* Those with a history of surgical treatment for the temporomandibular joint,
* Those with a history of allergy to any of the agents used in the treatment process,
* Those who use drugs that affect the musculoskeletal system, and
* Pregnant patients will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients with the history of limited mouth opening and TMJ arthralgia
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Maximum Amount of Mouth Opening | Measurements will be conducted at five time points, from enrollment through the 6-month follow-up period: (1) pre-arthrocentesis, (2) postoperative 1st week, (3) postoperative 1st month, (4) postoperative 3rd month, and (5) postoperative 6th month.
  For mouth opening measurement, the distance between the incisal edges of the lower and upper first incisors will be measured using a digital caliper and will be recorded in millimeters at the end of each examination. In patients with missing teeth, the teeth on the left side will be used for the measurement. In order to determine the amount of movement of the lower jaw in the lateral direction, patients will be asked to shift their lower jaws to the right and left. The amount of displacement of the midline of the lower jaw teeth relative to the midline of the upper jaw teeth will be measured with a digital caliper. The distances obtained will be recorded in millimeters at the end of each examination.
Pain Intensity | Measurements will be conducted at five time points, from enrollment through the 6-month follow-up period: (1) pre-arthrocentesis, (2) postoperative 1st week, (3) postoperative 1st month, (4) postoperative 3rd month, and (5) postoperative 6th month.
  A visual analog scale (VAS) will be used to measure pain intensity. The scale consists of a 10-centimeter straight line, with '0' at the starting point indicating no pain and '10' at the endpoint representing the highest pain level tolerable. During each examination session, individuals will mark the point on the line that corresponds to their pain intensity. The distance from the '0' point to the marked position will be measured in centimeters, with greater distances indicating higher pain intensity.

SECONDARY OUTCOMES:
Jaw Function Limitation | Measurements will be conducted at five time points, from enrollment through the 6-month follow-up period: (1) pre-arthrocentesis, (2) postoperative 1st week, (3) postoperative 1st month, (4) postoperative 3rd month, and (5) postoperative 6th month.
  The Jaw Function Limitation Scale (JFLS-20) will be administered to patients during all examination sessions using a standardized form. This scale assesses the extent to which daily activities are restricted by TMD symptoms. It includes 20 jaw functions, each scored by the patient on a scale from 0 to 10, where '0' indicates no impact and '10' indicates extreme difficulty performing the function due to TMD. The individual scores are summed to calculate a total score, with higher scores indicating greater limitations in jaw function.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Güngör, Prof Dr, Study Director — Uşak University
Locations (1):
- Uşak University, Faculty of Dentistry, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available upon request from the corresponding researcher following the publication of the study.

REFERENCES:
- [Background] Lindfors E, Arima T, Baad-Hansen L, Bakke M, De Laat A, Giannakopoulos NN, Glaros A, Guimaraes AS, Johansson A, Le Bell Y, Lobbezoo F, Michelotti A, Muller F, Ohrbach R, Wanman A, Magnusson T, Ernberg M. Jaw Exercises in the Treatment of Temporomandibular Disorders-An International Modified Delphi Study. J Oral Facial Pain Headache. 2019 Fall;33(4):389-398. doi: 10.11607/ofph.2359. Epub 2019 Jun 24. PMID 31247061
- [Background] Hosgor H, Bas B, Celenk C. A comparison of the outcomes of four minimally invasive treatment methods for anterior disc displacement of the temporomandibular joint. Int J Oral Maxillofac Surg. 2017 Nov;46(11):1403-1410. doi: 10.1016/j.ijom.2017.05.010. Epub 2017 Jun 9. PMID 28602569
- [Background] Bas B, Kazan D, Kutuk N, Gurbanov V. The Effect of Exercise on Range of Movement and Pain After Temporomandibular Joint Arthrocentesis. J Oral Maxillofac Surg. 2018 Jun;76(6):1181-1186. doi: 10.1016/j.joms.2018.01.003. Epub 2018 Jan 12. PMID 29406255